CLINICAL TRIAL: NCT01853202
Title: EXercise Training for the Prevention of Cancer Thrombosis (EXPECT) Pilot Trial
Acronym: EXPECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Susan Lakoski, Assistant Professor, University of Vermont College of Medicine, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VCC 1220
Record Dates: First submitted 2013-05-09; First posted 2013-05-14 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Cancer Thrombosis
Keywords: Cancer; Chemotherapy; Thrombosis; Prevention; Exercise
MeSH Terms: conditions — Neoplasms; Thrombosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 - Supervised aerobic exercise training (Experimental): This group will participate in 3 supervised exercise sessions/week at an intensity of 50%-70% of the individually determined VO2max between 30-45 min/session for 12 weeks. The aerobic training intervention will closely mimic the standard exercise-based guidelines adopted in cardiac rehabilitation. All intervention sessions will be performed in a supervised setting with one-on-one supervision by an American College of Sports Medicine-certified exercise physiologist. Aerobic exercise training will be prescribed based on the guiding ACSM principles with the aim of improving VO2max. Walking was chosen because it is the preferred mode of exercise training in cancer patients.
  Interventions: Behavioral: Supervised aerobic exercise training
- Group 2 (No Intervention): The 12-week program will consist of monthly phone contacts to check in with patient and review their exercise log entries for that month in order to capture physical activity done outside of the intervention setting.

INTERVENTIONS:
Behavioral: Supervised aerobic exercise training
  Arms: Group 1 - Supervised aerobic exercise training

SUMMARY:
Patients with lymphoma or cancer who are receiving chemotherapy in the outpatient setting are at risk for blood clots which form in the veins. The occurrence of blood clots has major implications on personal health including the need for blood thinners and monitoring, potential bleeding, and complications related to blood clots on cardiovascular health. The goal of this study is to determine whether aerobic exercise training is a therapeutic strategy to offset risk of blood clots and improve quality of life among cancer patients during chemotherapy.

DETAILED DESCRIPTION:
Activation of the blood coagulation system is a common manifestation in cancer associated with premature death from venous thromboembolism (VTE).(1-5) Ambulatory cancer patients undergoing chemotherapy for lymphoma or cancers such as lung, ovarian, stomach, bladder, and pancreas confer a 12.6% absolute rate of VTE at 1-year compared to similarly age-sex matched controls, with nearly 50% of VTE events occurring within the first 3 months of treatment.(6) Further, cancer patients who develop VTE have a 2.5-fold higher mortality risk compared to cancer patients who do not experience a VTE.(3) Therapies to offset VTE risk, such as low-molecular weight heparin or vitamin K antagonists, are not currently recommended by the American Society of Clinical Oncology Guidelines secondary to the lack of robust clinical trial data, potential bleeding, and need for monitoring and dose adjustment.(7) As such, alternative strategies to prevent VTE during chemotherapy without adding further toxicity are urgently required.

The investigators hypothesize aerobic exercise training is a therapeutic strategy to mitigate VTE risk among ambulatory cancer patients undergoing chemotherapy. Aerobic exercise training at moderate intensity has favorable effects on coagulation factors and reduces risk of VTE in healthy populations.(8-11) To date, no studies have determined whether exercise training has favorable impact on coagulation factors implicated in VTE risk. Furthermore, there is a lack of data regarding the impact of exercise training on functional performance and patient-reported outcomes among ambulatory cancer patients during chemotherapy. The focus of this grant application is to establish whether aerobic exercise training is as a potential modality to prevent VTE in ambulatory lymphoma and cancer patients during chemotherapy.

To this end, investigators propose the EXercise Training for the PrEvention of Cancer Thrombosis (EXPECT) Pilot trial, a two-arm randomized controlled trial (RCT) comparing aerobic exercise training (three supervised treadmill sessions per week on nonconsecutive days for 12 weeks at moderate intensity (50-70% of baseline VO2max)), versus control among 54 subjects (27/group). Patients with high risk VTE malignancies receiving chemotherapy in the ambulatory setting will be the focus of recruitment.(2, 6, 12) The primary endpoint will be change in thrombin generation,(13) as well as other established VTE risk markers in cancer.(14, 15) We will also assess relationships between exercise training and factor Xa generation, a key modulator of thrombosis and a novel therapeutic target for VTE prevention.(16, 17)

Design and Procedures: Potential participants will be identified and screened for eligibility by the study clinical research coordinator via medical record review of candidates scheduled to initiate chemotherapy at the Vermont Cancer Center. After obtaining written consent, all participants will complete the following baseline assessments: (1) fasting blood draw and (2) cardiopulmonary exercise test (CPET). Blood draws and CPET baseline assessments will be repeated at the end of the 12 week intervention.

Group (Randomization): Participants will be randomly allocated, on an individual basis, to one of the two study groups prior to the initiation of chemotherapy. Randomly allocated participants will remain in the same group for the remainder of the study (i.e., no cross-over). Randomization will be stratified by cancer type to ensure balance of types between groups.

Exercise Intervention:

All participants will agree to participate in exercise testing, exercise logging, blood draws, and surveys pre and post intervention. The intervention, depending on randomization, will include:

Group 1 - The goal of all AT groups is 3 supervised exercise sessions/week at an intensity of 50%-70% of the individually determined VO2max between 30-45 min/session for 12 weeks. The aerobic training intervention will closely mimic the standard exercise-based guidelines adopted in cardiac rehabilitation. All intervention sessions will be performed in a supervised setting with one-on-one supervision by an American College of Sports Medicine-certified exercise physiologist. Aerobic exercise training will be prescribed based on the guiding ACSM principles with the aim of improving VO2max. Walking was chosen because it is the preferred mode of exercise training in cancer patients.(51) Group 2 - Control: The 12-week program will consist of monthly phone contacts to check in with patient and review their exercise log entries for that month in order to capture physical activity done outside of the intervention setting.

Study Endpoints:

Markers of VTE Risk: Investigators will measure the following markers of VTE risk: thrombin, FXa, F 1+2, TAT, D-Dimer, vWF, soluble P-selectin, and C-reactive protein. Samples will be processed in the clinic with attention to issues related to coagulation activation, and plasma and serum will be stored at -80 degrees C in our laboratory.

Functional Capacity: VO2peak: To determine VO2peak, an incremental treadmill test (modified Balke protocol) with 12-lead ECG monitoring (Mortara) will be performed by ACSM-certified exercise physiologists. Expired gases will be analyzed continuously by a metabolic measurement system (Sensormedics Vmax 29c). Physical Functioning will also include both subjective (i.e., SF-36) assessment as well as a 6-min walk distance test as described previously.(55) Fatigue: The Fatigue Symptom Inventory (FSI) has been tested in several cancer patient populations and will be used to assess fatigue(56) Anxiety and depression will be assessed using The Medical Outcomes Study, Short Form Health Survey (SF-36). This is a widely used and validated instrument to assess general functional and health related quality of life.(58) The SF-36 is a 36 item instrument containing eight individual scales measuring the following domains: physical functioning, role physical, bodily pain, social functioning, mental health, vitality, role emotional and general health perceptions.

Exercise Experience: Individuals experience with exercise predicts participation in exercise interventions.

Exercise Self-Efficacy: Self-efficacy refers to one's belief that he/she can successfully complete a given activity.(59) Adherence will be evaluated by assessing the rates of study eligibility, acceptance, and overall accrual.

Safety will be evaluated by the type and prevalence of adverse events during exercise-related assessments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lymphoma or cancer
* Beginning chemotherapy regimen
* Patient self-report of ability to walk 10 minutes without interruption or pain
* Age >18 and <80
* Willingness to participate in the oncology rehabilitation program at Tilley Drive South Burlington

Exclusion Criteria:

* Presence or history of DVT or PE prior to entry
* Antithrombotic therapy including warfarin, dabigatran, low molecular weight heparin or unfractionated heparin which will alter levels of hemostatic factors (Off Lovenox 48 hours before first study blood draw)
* Medical condition that alters ability to walk for exercise

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Thrombin Generation | 12 weeks
  The primary endpoint will be thrombin generation, a marker of VTE risk in cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Susan G Lakoski, MD, Principal Investigator — University of Vermont
Locations (1):
- Fletcher Allen Healthcare, Burlington, Vermont, United States

REFERENCES:
- [Background] Khorana AA, Francis CW, Culakova E, Kuderer NM, Lyman GH. Thromboembolism is a leading cause of death in cancer patients receiving outpatient chemotherapy. J Thromb Haemost. 2007 Mar;5(3):632-4. doi: 10.1111/j.1538-7836.2007.02374.x. No abstract available. PMID 17319909
- [Background] Chew HK, Wun T, Harvey D, Zhou H, White RH. Incidence of venous thromboembolism and its effect on survival among patients with common cancers. Arch Intern Med. 2006 Feb 27;166(4):458-64. doi: 10.1001/archinte.166.4.458. PMID 16505267
- [Background] Levitan N, Dowlati A, Remick SC, Tahsildar HI, Sivinski LD, Beyth R, Rimm AA. Rates of initial and recurrent thromboembolic disease among patients with malignancy versus those without malignancy. Risk analysis using Medicare claims data. Medicine (Baltimore). 1999 Sep;78(5):285-91. doi: 10.1097/00005792-199909000-00001. PMID 10499070
- [Background] Flinterman LE, van Hylckama Vlieg A, Cannegieter SC, Rosendaal FR. Long-term survival in a large cohort of patients with venous thrombosis: incidence and predictors. PLoS Med. 2012 Jan;9(1):e1001155. doi: 10.1371/journal.pmed.1001155. Epub 2012 Jan 10. PMID 22253578
- [Background] Sorensen HT, Mellemkjaer L, Olsen JH, Baron JA. Prognosis of cancers associated with venous thromboembolism. N Engl J Med. 2000 Dec 21;343(25):1846-50. doi: 10.1056/NEJM200012213432504. PMID 11117976
- [Background] Khorana AA, Dalal M, Lin J, Connolly GC. Incidence and predictors of venous thromboembolism (VTE) among ambulatory high-risk cancer patients undergoing chemotherapy in the United States. Cancer. 2013 Feb 1;119(3):648-55. doi: 10.1002/cncr.27772. Epub 2012 Aug 14. PMID 22893596
- [Background] Lyman GH, Khorana AA, Falanga A, Clarke-Pearson D, Flowers C, Jahanzeb M, Kakkar A, Kuderer NM, Levine MN, Liebman H, Mendelson D, Raskob G, Somerfield MR, Thodiyil P, Trent D, Francis CW; American Society of Clinical Oncology. American Society of Clinical Oncology guideline: recommendations for venous thromboembolism prophylaxis and treatment in patients with cancer. J Clin Oncol. 2007 Dec 1;25(34):5490-505. doi: 10.1200/JCO.2007.14.1283. Epub 2007 Oct 29. PMID 17968019
- [Background] Wang JS. Exercise prescription and thrombogenesis. J Biomed Sci. 2006 Nov;13(6):753-61. doi: 10.1007/s11373-006-9105-7. Epub 2006 Aug 24. PMID 16933027
- [Background] Lee KW, Lip GY. Effects of lifestyle on hemostasis, fibrinolysis, and platelet reactivity: a systematic review. Arch Intern Med. 2003 Oct 27;163(19):2368-92. doi: 10.1001/archinte.163.19.2368. PMID 14581258
- [Background] van Stralen KJ, Le Cessie S, Rosendaal FR, Doggen CJ. Regular sports activities decrease the risk of venous thrombosis. J Thromb Haemost. 2007 Nov;5(11):2186-92. doi: 10.1111/j.1538-7836.2007.02732.x. Epub 2007 Aug 14. PMID 17697136
- [Background] Rauramaa R, Li G, Vaisanen SB. Dose-response and coagulation and hemostatic factors. Med Sci Sports Exerc. 2001 Jun;33(6 Suppl):S516-20; discussion S528-9. doi: 10.1097/00005768-200106001-00022. PMID 11427778
- [Background] Khorana AA, Kuderer NM, Culakova E, Lyman GH, Francis CW. Development and validation of a predictive model for chemotherapy-associated thrombosis. Blood. 2008 May 15;111(10):4902-7. doi: 10.1182/blood-2007-10-116327. Epub 2008 Jan 23. PMID 18216292
- [Background] Ay C, Dunkler D, Simanek R, Thaler J, Koder S, Marosi C, Zielinski C, Pabinger I. Prediction of venous thromboembolism in patients with cancer by measuring thrombin generation: results from the Vienna Cancer and Thrombosis Study. J Clin Oncol. 2011 May 20;29(15):2099-103. doi: 10.1200/JCO.2010.32.8294. Epub 2011 Apr 4. PMID 21464402
- [Background] Ay C, Vormittag R, Dunkler D, Simanek R, Chiriac AL, Drach J, Quehenberger P, Wagner O, Zielinski C, Pabinger I. D-dimer and prothrombin fragment 1 + 2 predict venous thromboembolism in patients with cancer: results from the Vienna Cancer and Thrombosis Study. J Clin Oncol. 2009 Sep 1;27(25):4124-9. doi: 10.1200/JCO.2008.21.7752. Epub 2009 Jul 27. PMID 19636003
- [Background] Connolly GC, Khorana AA. Risk stratification for cancer-associated venous thromboembolism. Best Pract Res Clin Haematol. 2009 Mar;22(1):35-47. doi: 10.1016/j.beha.2008.12.006. PMID 19285271
- [Background] Ansell J. Factor Xa or thrombin: is factor Xa a better target? J Thromb Haemost. 2007 Jul;5 Suppl 1:60-4. doi: 10.1111/j.1538-7836.2007.02473.x. PMID 17635710
- [Background] Gomez-Outes A, Terleira-Fernandez AI, Suarez-Gea ML, Vargas-Castrillon E. Dabigatran, rivaroxaban, or apixaban versus enoxaparin for thromboprophylaxis after total hip or knee replacement: systematic review, meta-analysis, and indirect treatment comparisons. BMJ. 2012 Jun 14;344:e3675. doi: 10.1136/bmj.e3675. PMID 22700784
- [Background] Heit JA, Silverstein MD, Mohr DN, Petterson TM, O'Fallon WM, Melton LJ 3rd. Risk factors for deep vein thrombosis and pulmonary embolism: a population-based case-control study. Arch Intern Med. 2000 Mar 27;160(6):809-15. doi: 10.1001/archinte.160.6.809. PMID 10737280
- [Background] Silverstein MD, Heit JA, Mohr DN, Petterson TM, O'Fallon WM, Melton LJ 3rd. Trends in the incidence of deep vein thrombosis and pulmonary embolism: a 25-year population-based study. Arch Intern Med. 1998 Mar 23;158(6):585-93. doi: 10.1001/archinte.158.6.585. PMID 9521222
- [Background] Agnelli G, George DJ, Kakkar AK, Fisher W, Lassen MR, Mismetti P, Mouret P, Chaudhari U, Lawson F, Turpie AG; SAVE-ONCO Investigators. Semuloparin for thromboprophylaxis in patients receiving chemotherapy for cancer. N Engl J Med. 2012 Feb 16;366(7):601-9. doi: 10.1056/NEJMoa1108898. PMID 22335737
- [Background] Akl EA, Vasireddi SR, Gunukula S, Yosuico VE, Barba M, Terrenato I, Sperati F, Schunemann H. Oral anticoagulation in patients with cancer who have no therapeutic or prophylactic indication for anticoagulation. Cochrane Database Syst Rev. 2010 Dec 8;(12):CD006466. doi: 10.1002/14651858.CD006466.pub2. PMID 21154368
- [Background] Kahn SR, Lim W, Dunn AS, Cushman M, Dentali F, Akl EA, Cook DJ, Balekian AA, Klein RC, Le H, Schulman S, Murad MH. Prevention of VTE in nonsurgical patients: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e195S-e226S. doi: 10.1378/chest.11-2296. PMID 22315261
- [Background] Lockard MM, Gopinathannair R, Paton CM, Phares DA, Hagberg JM. Exercise training-induced changes in coagulation factors in older adults. Med Sci Sports Exerc. 2007 Apr;39(4):587-92. doi: 10.1249/mss.0b013e31802eff4b. PMID 17414794
- [Background] Wannamethee SG, Lowe GD, Whincup PH, Rumley A, Walker M, Lennon L. Physical activity and hemostatic and inflammatory variables in elderly men. Circulation. 2002 Apr 16;105(15):1785-90. doi: 10.1161/hc1502.107117. PMID 11956120
- [Background] Wang JS, Li YS, Chen JC, Chen YW. Effects of exercise training and deconditioning on platelet aggregation induced by alternating shear stress in men. Arterioscler Thromb Vasc Biol. 2005 Feb;25(2):454-60. doi: 10.1161/01.ATV.0000151987.04607.24. Epub 2004 Nov 29. PMID 15569820
- [Background] Lindqvist PG, Epstein E, Olsson H. The relationship between lifestyle factors and venous thromboembolism among women: a report from the MISS study. Br J Haematol. 2009 Jan;144(2):234-40. doi: 10.1111/j.1365-2141.2008.07460.x. Epub 2008 Nov 19. PMID 19036105
- [Background] Jones LW, Courneya KS, Mackey JR, Muss HB, Pituskin EN, Scott JM, Hornsby WE, Coan AD, Herndon JE 2nd, Douglas PS, Haykowsky M. Cardiopulmonary function and age-related decline across the breast cancer survivorship continuum. J Clin Oncol. 2012 Jul 10;30(20):2530-7. doi: 10.1200/JCO.2011.39.9014. Epub 2012 May 21. PMID 22614980
- [Background] Wang T, Nelson RA, Bogardus A, Grannis FW Jr. Five-year lung cancer survival: which advanced stage nonsmall cell lung cancer patients attain long-term survival? Cancer. 2010 Mar 15;116(6):1518-25. doi: 10.1002/cncr.24871. PMID 20108308
- [Background] Patnaik SK, Kannisto E, Mallick R, Yendamuri S. Overexpression of the lung cancer-prognostic miR-146b microRNAs has a minimal and negative effect on the malignant phenotype of A549 lung cancer cells. PLoS One. 2011;6(7):e22379. doi: 10.1371/journal.pone.0022379. Epub 2011 Jul 18. PMID 21789255
- [Background] Patnaik JL, Byers T, Diguiseppi C, Denberg TD, Dabelea D. The influence of comorbidities on overall survival among older women diagnosed with breast cancer. J Natl Cancer Inst. 2011 Jul 20;103(14):1101-11. doi: 10.1093/jnci/djr188. Epub 2011 Jun 30. PMID 21719777
- [Background] Wei S, Pan Z, Siegal GP, Winokur TS, Carroll AJ, Jhala D. Complex analysis of a recurrent pleomorphic hyalinizing angiectatic tumor of soft parts. Hum Pathol. 2012 Jan;43(1):121-6. doi: 10.1016/j.humpath.2011.02.023. Epub 2011 Jul 5. PMID 21733556
- [Background] Schmitz KH, Courneya KS, Matthews C, Demark-Wahnefried W, Galvao DA, Pinto BM, Irwin ML, Wolin KY, Segal RJ, Lucia A, Schneider CM, von Gruenigen VE, Schwartz AL; American College of Sports Medicine. American College of Sports Medicine roundtable on exercise guidelines for cancer survivors. Med Sci Sports Exerc. 2010 Jul;42(7):1409-26. doi: 10.1249/MSS.0b013e3181e0c112. PMID 20559064
- [Background] Evenson KR, Stevens J, Thomas R, Cai J. Effect of cardiorespiratory fitness on mortality among hypertensive and normotensive women and men. Epidemiology. 2004 Sep;15(5):565-72. doi: 10.1097/01.ede.0000129527.53181.c8. PMID 15308956
- [Background] Knols R, Aaronson NK, Uebelhart D, Fransen J, Aufdemkampe G. Physical exercise in cancer patients during and after medical treatment: a systematic review of randomized and controlled clinical trials. J Clin Oncol. 2005 Jun 1;23(16):3830-42. doi: 10.1200/JCO.2005.02.148. PMID 15923576
- [Background] Galvao DA, Newton RU. Review of exercise intervention studies in cancer patients. J Clin Oncol. 2005 Feb 1;23(4):899-909. doi: 10.1200/JCO.2005.06.085. PMID 15681536
- [Background] Zwicker JI, Furie BC, Furie B. Cancer-associated thrombosis. Crit Rev Oncol Hematol. 2007 May;62(2):126-36. doi: 10.1016/j.critrevonc.2007.01.001. Epub 2007 Feb 12. PMID 17293122
- [Background] Caine GJ, Stonelake PS, Lip GY, Kehoe ST. The hypercoagulable state of malignancy: pathogenesis and current debate. Neoplasia. 2002 Nov-Dec;4(6):465-73. doi: 10.1038/sj.neo.7900263. PMID 12407439
- [Background] Rickles FR, Falanga A. Molecular basis for the relationship between thrombosis and cancer. Thromb Res. 2001 Jun 15;102(6):V215-24. doi: 10.1016/s0049-3848(01)00285-7. PMID 11516455
- [Background] Rickles FR, Patierno S, Fernandez PM. Tissue factor, thrombin, and cancer. Chest. 2003 Sep;124(3 Suppl):58S-68S. doi: 10.1378/chest.124.3_suppl.58s. PMID 12970125
- [Background] Butenas S, Mann KG. Blood coagulation. Biochemistry (Mosc). 2002 Jan;67(1):3-12. doi: 10.1023/a:1013985911759. PMID 11841335
- [Background] Butenas S, van 't Veer C, Mann KG. Evaluation of the initiation phase of blood coagulation using ultrasensitive assays for serine proteases. J Biol Chem. 1997 Aug 22;272(34):21527-33. doi: 10.1074/jbc.272.34.21527. PMID 9261172
- [Background] Brummel-Ziedins K, Undas A, Orfeo T, Gissel M, Butenas S, Zmudka K, Mann KG. Thrombin generation in acute coronary syndrome and stable coronary artery disease: dependence on plasma factor composition. J Thromb Haemost. 2008 Jan;6(1):104-10. doi: 10.1111/j.1538-7836.2007.02799.x. Epub 2007 Oct 15. PMID 17944993
- [Background] Gissel M, Undas A, Slowik A, Mann KG, Brummel-Ziedins KE. Plasma factor and inhibitor composition contributes to thrombin generation dynamics in patients with acute or previous cerebrovascular events. Thromb Res. 2010 Oct;126(4):262-9. doi: 10.1016/j.thromres.2010.07.002. Epub 2010 Aug 14. PMID 20709367
- [Background] Brummel-Ziedins K, Vossen CY, Rosendaal FR, Umezaki K, Mann KG. The plasma hemostatic proteome: thrombin generation in healthy individuals. J Thromb Haemost. 2005 Jul;3(7):1472-81. doi: 10.1111/j.1538-7836.2005.01249.x. PMID 15978105
- [Background] Brummel KE, Paradis SG, Butenas S, Mann KG. Thrombin functions during tissue factor-induced blood coagulation. Blood. 2002 Jul 1;100(1):148-52. doi: 10.1182/blood.v100.1.148. PMID 12070020
- [Background] Baglin T. The measurement and application of thrombin generation. Br J Haematol. 2005 Sep;130(5):653-61. doi: 10.1111/j.1365-2141.2005.05612.x. PMID 16115120
- [Background] Goldenberg N, Kahn SR, Solymoss S. Markers of coagulation and angiogenesis in cancer-associated venous thromboembolism. J Clin Oncol. 2003 Nov 15;21(22):4194-9. doi: 10.1200/JCO.2003.05.165. PMID 14615447
- [Background] Brummel-Ziedins KE, Orfeo T, Gissel M, Mann KG, Rosendaal FR. Factor Xa generation by computational modeling: an additional discriminator to thrombin generation evaluation. PLoS One. 2012;7(1):e29178. doi: 10.1371/journal.pone.0029178. Epub 2012 Jan 11. PMID 22247769
- [Background] Nalluri SR, Chu D, Keresztes R, Zhu X, Wu S. Risk of venous thromboembolism with the angiogenesis inhibitor bevacizumab in cancer patients: a meta-analysis. JAMA. 2008 Nov 19;300(19):2277-85. doi: 10.1001/jama.2008.656. PMID 19017914
- [Background] Jones LW, Eves ND, Haykowsky M, Joy AA, Douglas PS. Cardiorespiratory exercise testing in clinical oncology research: systematic review and practice recommendations. Lancet Oncol. 2008 Aug;9(8):757-65. doi: 10.1016/S1470-2045(08)70195-5. PMID 18672211
- [Background] Cushman M, Cornell ES, Howard PR, Bovill EG, Tracy RP. Laboratory methods and quality assurance in the Cardiovascular Health Study. Clin Chem. 1995 Feb;41(2):264-70. PMID 7874780
- [Background] Hockin MF, Jones KC, Everse SJ, Mann KG. A model for the stoichiometric regulation of blood coagulation. J Biol Chem. 2002 May 24;277(21):18322-33. doi: 10.1074/jbc.M201173200. Epub 2002 Mar 13. PMID 11893748
- [Background] Butenas S, Orfeo T, Gissel MT, Brummel KE, Mann KG. The significance of circulating factor IXa in blood. J Biol Chem. 2004 May 28;279(22):22875-82. doi: 10.1074/jbc.M400531200. Epub 2004 Mar 23. PMID 15039440
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Hann DM, Jacobsen PB, Azzarello LM, Martin SC, Curran SL, Fields KK, Greenberg H, Lyman G. Measurement of fatigue in cancer patients: development and validation of the Fatigue Symptom Inventory. Qual Life Res. 1998 May;7(4):301-10. doi: 10.1023/a:1024929829627. PMID 9610214
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Marcus BH, Selby VC, Niaura RS, Rossi JS. Self-efficacy and the stages of exercise behavior change. Res Q Exerc Sport. 1992 Mar;63(1):60-6. doi: 10.1080/02701367.1992.10607557. PMID 1574662
- [Background] Ay C, Haselbock J, Laczkovics C, Koder S, Pabinger I. Thrombin generation in patients with a bleeding tendency of unknown origin. Ann Hematol. 2011 Sep;90(9):1099-104. doi: 10.1007/s00277-011-1201-8. Epub 2011 Feb 26. PMID 21359651
- [Background] Poerwanto S, Stevenson M, de Klerk N. Infant mortality and family welfare: policy implications for Indonesia. J Epidemiol Community Health. 2003 Jul;57(7):493-8. doi: 10.1136/jech.57.7.493. PMID 12821691
- [Background] Jones LW, Eves ND, Mackey JR, Peddle CJ, Haykowsky M, Joy AA, Courneya KS, Tankel K, Spratlin J, Reiman T. Safety and feasibility of cardiopulmonary exercise testing in patients with advanced cancer. Lung Cancer. 2007 Feb;55(2):225-32. doi: 10.1016/j.lungcan.2006.10.006. Epub 2006 Nov 17. PMID 17113185
- [Background] Jones LW, Eves ND, Peterson BL, Garst J, Crawford J, West MJ, Mabe S, Harpole D, Kraus WE, Douglas PS. Safety and feasibility of aerobic training on cardiopulmonary function and quality of life in postsurgical nonsmall cell lung cancer patients: a pilot study. Cancer. 2008 Dec 15;113(12):3430-9. doi: 10.1002/cncr.23967. PMID 18988290